CLINICAL TRIAL: NCT03850093
Title: Preoperative Gabapentin Versus Bisoprolol for Intraoperative Hemodynamic and Surgical Field Optimization During Endoscopic Sinus Surgery
Brief Title: Preoperative Gabapentin Versus Bisoprolol for Hemodynamic Optimization During Sinus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, abeer M. elnakera, assistant professor of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZU-IRB 2139-24-5-2015
Record Dates: First submitted 2019-02-18; First posted 2019-02-21 (Actual); Results first posted 2019-08-12 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Blood Pressure
Keywords: gabapentin; bisoprolol; hemodynamic; surgical field
MeSH Terms: interventions — Bisoprolol; Vitamins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- gabapentin (Active Comparator): gabapentin 1200 mg was given to patients of gabapentin group 2 hours preoperative
  Interventions: Drug: Gabapentin1200 mg
- bisoprolol (Active Comparator): bisoprolol 2.5 mg was given to patients of bisoprolol group 2 hours preoperative
  Interventions: Drug: bisoprolol 2.5mg
- control (Placebo Comparator): placebo was given to patients of control group 2 hours preoperative
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Gabapentin1200 mg — patients received 1200mg gabapentin 2 hrs preoperative
  Other Names: gaptin
  Arms: gabapentin
Drug: bisoprolol 2.5mg — patients received 2.5mg bisoprolol 2 hrs preoperative
  Other Names: concor
  Arms: bisoprolol
Drug: placebo — patients received oral placebo 2 hrs preoperative
  Other Names: vitamins
  Arms: control

SUMMARY:
the current study hypothesized that Gabapentin can be effective as Bisoprolol in reduction of intraoperative bleeding, improving the operative's field visibility and increase the surgeon satisfaction via optimization of blood pressure and heart rate .

A prospective randomized double blinded controlled study. Eligible patients were randomized according to random list generated software and allocated into 3 equal and matched groups (15 patients in each group):-

* Group G: gabapentin group in which Patients were premedicated with oral gabapentin 1200 mg (Conventin 400mg; Evapharm) with sips of water, 2 hours before induction of anesthesia.
* Group B: bisoprolol group in which Patients were premedicated with oral bisoprolol 2.5 mg ( Concor 2.5mg ; Merck/Amoun ) with sips of water, 2 hours before induction of anesthesia.
* Group C: control group in which Patients were premedicated with oral placebo with sips of water, 2 hours before induction of anesthesia.

DETAILED DESCRIPTION:
Hypothesis:

Gabapentin can be effective as Bisoprolol in reduction of intraoperative bleeding, improving the operative's field visibility and increase the surgeon satisfaction via optimization of blood pressure and heart rate.

Objectives Compare the effect of preoperative Gabapentin with Bisoprolol on hemodynamics, surgical field optimization during endoscopic nasal surgeries.

Technical design:

A) Site of study :

The study was conducted at Anesthesia and Surgical intensive care and Otorhinolaryngology departments, faculty of medicine, Zagazig University.

B) Sample Size :

According to 80% power of the study, 95% CI and calculated volume of blood loss 200±40 ml and 150±55ml on Gabapentin (22) and Bisoprolol (15) premedication respectively, the estimated Sample size was 54 patients (open EPI) , 63 patients were included in the study to compensate for drop out.

Randomization was carried out on 63 patients to compensate for drop out . All planned ESS procedures was managed by the same anesthetist and surgeon who were blinded to the used study's premedication. The surgeon was blinded to the monitor recording the hemodynamic variables.

All patients had been preoperatively evaluated according to standard local protocol. Preoperative surgical preparation and proper management of infection were confirmed to every patient.

Patient was premedicated by IV ranitidine 50 mg, midazolam 0.05 mg/kg and atropine 20µg/kg immediately before admission to the operating room.

On admission to the operating room, Standard monitoring included 5 leads ECG, non-invasive blood pressure, Pulse Oximetry and End-tidal carbon dioxide (ETCO2) trace were applied (B40i Monitor - GE Healthcare, Finland).

Anesthesia was induced with IV propofol 2 mg/kg and fentanyl 1 µg/kg was given for analgesia. Cisatracurium 0.15 mg/kg IV was given to facilitate direct laryngoscopy and orotracheal intubation. The patient was ventilated at tidal volume 6-8mL/kg and respiratory rate that achieved ETCO2 of 30-35 mmHg. Oropharyngeal pack was inserted.

Anesthesia was maintained by isoflurane based on MAC 1.2 % until a steady state of anesthesia was achieved (defined as a state of anesthesia when no changes in hemodynamic variables take place for at least 10 min). An increase of ≥ 20% of basal value in both HR and MAP was treated with increasing the concentration of isoflurane by 0.5% and increments of fentanyl 1 μg/kg. Muscle relaxation was confirmed by cisatracurium 0.03mg/kg every 20 mins. IV lactated ringer solution was infused at approximately 6ml/kg/hr till the end of the procedure.

All patients were positioned supine and the bed-head of the surgical table was raised by 30° to improve venous drainage.

Before the beginning of surgical procedure, well wrung out cotton pledgets soaked with 4 ml of 2% lignocaine with 1:200,000 adrenaline were topically applied to the nasal mucous membrane for 10 min (no infiltration).

Technique for hemodynamic optimization:

Target mean arterial pressure (MAP) was 60-70 mmHg during the surgical procedure to achieve Fromm and Boezaart category scale of 2 or 3 which is judged to be optimal for surgery (20).

If the MAP was still ˃70mmHg in spite of increasing isoflurane inhalation to 2.5%, nitroglycerine (1-10 μg/kg/min.) titrated to effect.

If the heart rate was more than 100 beats/ minute, propranolol was titrated 1-3 mg/hour to achieve target MAP.

If mean arterial pressure (MAP) decreased to less than 60 mm Hg, ephedrine in increments of 3 mg was given.

Withdrawal vasoactive agents:

After recording the surgeons' opinion regarding the surgical field and about 15 minutes before ending surgery, the infusion of any vasoactive medication (if used) was stopped and the anesthetic agent was decreased allowing HR and MAP to return to their basal value. If Hypotension (defined as SAP< 90mmHg and bradycardia less than 60 bpm) persisted, they was treated by ephedrine in increments of 3 mg .

On compilation of surgical procedure, anesthesia was discontinued and reversal of neuromuscular blockade was achieved using IV neostigmine 0.08 mg/kg and atropine 20µg/kg. After removal of oropharyngeal pack, oropharyngeal suction was performed. On the start of obeying commands, patients were extubated and shifted to recovery room.

Patients were discharged to the ward after reaching a score ≥ 9 on the Modified Aldrete Scoring System.

During postoperative period up to 6 hours, the patient was monitored for conscious level, oxygen saturation, heart rate and mean arterial blood pressure.

On ward admission, IM diclofenac sodium 75mg was given then every 12 hours. If the patient complained moderate to severe pain (VAS≥ 4) meperidine 25mg increments up to pain relief (maximum 100mg as a single dose) was given.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent functional endoscopic sinus surgery
* ability to swallow tablets

Exclusion Criteria:

* suspected difficult airway
* basal HR <60/min.
* chronic cardiovascular or cerebrovascular disease
* bronchial asthma or COPD
* DM
* bleeding disorders
* anemia (Hb level< 10 gm/dl)
* renal or hepatic insufficiency
* psychiatric disorders
* chronic treatment by BBs, gabapentin or drugs that affect coagulation
* acute nasal infection
* allergy/contraindications to any of the study's drugs.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abeer M. Elnakera, doctorate, Principal Investigator — faculty of medicine - Zagazig university; Ayman A. Hassan, doctorate, Study Chair — Zagazig University; Maram wagdy, Master, Study Chair — Zagazig University; Mohamed W. El-Anwar, doctorate, Study Chair — Zagazig University

IPD SHARING:
Plan to Share IPD: No
collective data sheet was available to all researchers during and after completing the study. individual patient records are available on request for all researchers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 66 patients who underwent endoscopic sinus surgery were eligible for the study
Groups:
- Gabapentin Group (Group G): 21 patients completed the study and were considered for statistical analysis
- Bisoprolol Group (Group B): 22 patients were allocated to group B, completed the study and were considered for statistical analysis
- Control Group (Group C): 17 patients completed the study and were considered for statistical analysis
Period: Overall Study
Arm/Group | Gabapentin Group (Group G) | Bisoprolol Group (Group B) | Control Group (Group C)
Started | 22 | 22 | 19
Completed | 21 | 22 | 17
Not Completed | 1 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: 63 patients were enrolled in the study. after 3 patients' withdrawal, 60 patients completed the study and considered for statistical analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Bisoprolol | Control | Total
Number analyzed (Participants) | 21 | 22 | 17 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (7.6) | 30.5 (6.6) | 28.6 (5.1) | 27.93 (6.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 6 | 23
  Male | 13 | 13 | 11 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
weight, continuous [Mean (Standard Deviation); unit: kilograms] — Population: patients' withdrawal from the study
  kilograms | 87.1 (1.1) | 87.9 (11.9) | 84.5 (11.5) | 85.62 (11.5)
indication for surgery, categorical) [Count of Participants; unit: Participants] — indication for surgery is either due to polyp or sinusitis Population: 3 patients were withdrawn from the study
  Participants
    polyp | 11 | 13 | 10 | 34
    sinusitis | 10 | 9 | 7 | 26
mean arterial blood pressure (MAP), continuous [Mean (Standard Deviation); unit: mmHg] — Population: 3 patients were withdrawn from the study
  mmHg | 96.6 (7.5) | 92.9 (7.4) | 88.2 (11.7) | 93.4 (9.7)
heart rate (HR), continuous [Mean (Standard Deviation); unit: beats/minute] — Population: 3 patients were withdrawn from the study
  beats/minute | 91.1 (11.6) | 82.9 (6.4) | 83.8 (14.8) | 86.7 (11.98)
side of surgery [Count of Participants; unit: Participants] — side of surgery is either bilateral or unilateral Population: 3 patients were withdrawn from the study
  Participants
    bilateral | 14 | 11 | 9 | 34
    unilateral | 7 | 11 | 8 | 26

OUTCOME MEASURES:

1. Primary Outcome: Changes in Surgical Field Visibility
Description: according to change in Fromm and Boezaart surgical field category scale ranging from 0 (no bleeding) to 5 (severe bleeding) where: 0 No Bleeding.
  1. Slight bleeding- no blood suctioning required.
  2. Slight bleeding- occasional blood suctioning required.
  3. Slight bleeding- frequent blood suctioning required, operative field is visible for some seconds after evacuation.
  4. Moderate bleeding- frequent blood suctioning required, operative field is only visible immediately after evacuation.
  5. Severe bleeding- constant blood suctioning required, bleeding appears faster than can be removed by suction .Surgery is hardly possible, and sometimes impossible.
Time Frame: scale was assessed by the surgeon every 15 minutes from the start of surgical procedure till the end
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Gabapentin | Bisoprolol | Control
Number analyzed (Participants) | 21 | 22 | 17
score on a scale
  15 minutes | 2 [2 to 3] | 2 [1 to 3] | 4 [3 to 4]
  30 minutes | 1 [1 to 3] | 1 [1 to 2] | 3 [2 to 4]
  45 minutes | 1 [0 to 2] | 1 [1 to 3] | 3 [2 to 3]
  60 minutes | 1 [0 to 1] | 1 [1 to 2] | 3 [3 to 4]
  75 minutes | 1 [1 to 2] | 1 [0 to 2] | 2 [2 to 3]
  90 minutes | 1 [0 to 2] | 0 [0 to 2] | 3 [2 to 3]
  105 minutes | 1 [0 to 2] | 0 [0 to 2] | 2 [2 to 3]

2. Primary Outcome: Blood Loss
Description: total intraoperative blood loss (mL)
Time Frame: at the end of surgery
Measure: Median (Full Range); unit: mL
Arm/Group | Gabapentin | Bisoprolol | Control
Number analyzed (Participants) | 21 | 22 | 17
mL | 20 [10 to 40] | 20 [10 to 30] | 80 [30 to 110]

3. Secondary Outcome: Heart Rate Change
Description: effect of intervention on the change of heart rate allover study period
Time Frame: were recorded before oral premedication (baseline), pre-induction, after induction of anesthesia, 1, 5, 10, 15 minutes after intubation and then every 15 minutes until the end of surgery
Measure: Mean (Standard Deviation); unit: beats/ minute
Arm/Group | Gabapentin | Bisoprolol | Control
Number analyzed (Participants) | 21 | 22 | 17
beats/ minute
  preinduction | 82.6 (10.4) | 73.1 (9.5) | 85.8 (16)
  after induction | 74.9 (11.8) | 67.8 (6.8) | 85.9 (16.7)
  1 minute after intubation | 83.3 (11.1) | 73.3 (9.4) | 96.2 (18.8)
  5 minutes after intubation | 77.1 (10) | 70.6 (8.8) | 89.3 (17.5)
  10 minutes after intubation | 75.4 (8.6) | 66.3 (5.4) | 87.8 (19.1)
  15 minutes after intubation | 74.7 (8.8) | 66.6 (5.8) | 90.2 (19.8)
  30 minutes after intubation | 73.4 (9.4) | 67.7 (4.9) | 85.8 (14.3)
  45 minutes after intubation | 75 (7.4) | 67.1 (4.2) | 80.1 (14.7)
  60 minutes after intubation | 75.3 (7.4) | 66.3 (4.8) | 87.3 (13.5)
  75 minutes after intubation | 75.7 (8.9) | 66 (4.3) | 84.5 (14.1)
  90 minutes after intubation | 72.7 (8.4) | 66.5 (3.4) | 88.1 (14.3)
  105 minutes after intubation | 75.7 (8.1) | 67.4 (5.7) | 97 (13.2)

4. Secondary Outcome: Mean Arterial Blood Pressure Change
Description: effect of intervention on the change of mean arterial blood pressure allover study period
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Gabapentin | Bisoprolol | Control
Number analyzed (Participants) | 21 | 22 | 17
mm Hg
  preinduction | 85.6 (6) | 86.4 (6.6) | 92.4 (9.8)
  after induction | 74.4 (6.9) | 72.3 (9.9) | 78.2 (9.1)
  1 minute after intubation | 80.6 (7.6) | 76.2 (12.9) | 92.2 (16.1)
  5 minutes after intubation | 70.7 (8.4) | 67.2 (7.8) | 78.6 (11.1)
  10 minutes after intubation | 66.4 (7.1) | 67.7 (10.4) | 76.5 (12.9)
  15 minutes after intubation | 65.4 (4.6) | 70.2 (8.8) | 74 (12.1)
  30 minutes after intubation | 64.4 (4.4) | 66.2 (6.8) | 66.6 (21.7)
  45 minutes after intubation | 63.3 (3.4) | 64.7 (6.6) | 64.6 (14.3)
  60 minutes after intubation | 61.9 (4.2) | 66.7 (4.8) | 69.9 (11.3)
  75 minutes after intubation | 62.5 (4.4) | 69.4 (8.4) | 67.7 (5.5)
  90 minutes after intubation | 63 (3.5) | 66.1 (4.7) | 62.7 (12.8)
  105 minutes after intubation | 63.1 (3) | 67.2 (7.7) | 70 (14.8)

5. Other Pre Specified Outcome: Surgeon Satisfaction (Categorical)
Description: surgeon satisfaction score where given 5 for very satisfied, 4 for satisfied, 3 for neutral, 2 for dissatisfied and 1 for very dissatisfied then number of satisfied (satisfaction score = 5) and disatisfied (satisfaction score less than 5) surgeons was compared between groups
Time Frame: at the end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Bisoprolol | Control
Number analyzed (Participants) | 21 | 22 | 17
Participants
  surgeon satisfaction achieved (score≥ 4) | 21 | 22 | 10
  surgeon satisfaction not achieved(score< 4) | 0 | 0 | 7

6. Other Pre Specified Outcome: Number of Patients Who Recieved Intraoperative IV Nitroglycerin During Operative Procedure
Description: need for additional intraoperative IV vasodilators (nitroglycerine
Time Frame: at the end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Bisoprolol | Control
Number analyzed (Participants) | 21 | 22 | 17
Participants | 0 | 0 | 5

7. Other Pre Specified Outcome: Number of Patients Who Recieved Intraoperative IV Propranolol During Operative Procedure
Description: the need for additional beta blockers (propranolol)
Time Frame: at the end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Bisoprolol | Control
Number analyzed (Participants) | 21 | 22 | 17
Participants | 0 | 0 | 1

8. Other Pre Specified Outcome: Number of Patients Who Recieve Both IV Nitroglycerin and Propranolol During Operative Procedure
Description: need for both IV nitroglycerine and propranolol intraoperatively
Time Frame: at the end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Bisoprolol | Control
Number analyzed (Participants) | 21 | 22 | 17
Participants | 0 | 0 | 6

9. Other Pre Specified Outcome: Visual Analogue Scale (VAS) for Postoperative Pain
Description: postoperative visual analogue score (VAS) for pain where 0 is no pain and 10 severe intolerable pain which was assessed
Time Frame: 1, 3 and 6 hrs. after recovery
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Visual Analogue Scale (VAS) for Postoperative Pain
Description: postoperative visual analogue score (VAS) for pain where 0 is no pain and 10 severe intolerable pain
Time Frame: 0n full recovery, 3 and 6 hrs. after recovery
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Gabapentin | Bisoprolol | Control
Number analyzed (Participants) | 21 | 22 | 17
score on a scale
  on full recovery | 2 [0 to 4] | 4 [3 to 5] | 5 [4 to 6]
  3hrs. after recovery | 1 [0 to 3] | 3 [2 to 4] | 4 [3 to 4]
  6hrs after recovery | 1 [0 to 3] | 3 [2 to 4] | 3 [2 to 4]

11. Other Pre Specified Outcome: Time to 1st Postoperative Rescue Analgesia
Description: time to 1st postoperative rescue analgesia (starting from administration of the studied drug)
Time Frame: on administration of 1st postoperative rescue analgesia
Measure: Median (Full Range); unit: minutes
Arm/Group | Gabapentin | Bisoprolol | Control
Number analyzed (Participants) | 21 | 22 | 17
minutes | 60 [0 to 90] | 30 [20 to 50] | 20 [0 to 30]

ADVERSE EVENTS:
Time Frame: intra-operative and up to 6 hours postoperative
Description: hypertension:MAP elevation by more than 20% from baseline value hypotension : systolic arterial pressure (SAP) less than 90 mmHg tachycardia : HR more than 90 beats/min bradycardia: HR less than 60 beats/min incidence of nausea and vomiting
Arm/Group | Gabapentin | Bisoprolol | Control
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/21 | 5/22 | 11/17
Other Adverse Events (participants affected / at risk) | 0/21 | 3/22 | 10/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gabapentin (N=21) | Bisoprolol (N=22) | Control (N=17)
hypotension (Cardiac disorders) | 0 | 1 | 7 — SAP less than 90 mmHg
bradycardia (Cardiac disorders) | 0 | 4 | 4 — HR less than 60 beats/min
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=21) | Bisoprolol (N=22) | Control (N=17)
hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 10 (20) — MAP elevation by more than 20% from baseline
tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 9 (18) — HR more than 90 beats/min
postoperative nausea (Gastrointestinal disorders) | 0 (0) | 3 (6) | 5 (10)
postoperative vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
agitation on recovery (Nervous system disorders) | 0 (0) | 0 (0) | 5 (5) — Richmond Agitation Sedation Scale (RASS) equal +2

LIMITATIONS AND CAVEATS:
small sample size, short study period (until 6 hrs. postoperatively) and unavailability of BIS index monitoring.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT03850093/SAP_000.pdf